CLINICAL TRIAL: NCT04151342
Title: CAnadian CAncers With Rare Molecular Alterations (CARMA) - Basket Real-world Observational Study (BROS)
Acronym: CARMA-BROS
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Takeda Canada, Inc. (Industry); Applied Health Research Centre (Other); Programs for Assessment of Technology in Health Research Institute (Other); AstraZeneca (Industry); Amgen (Industry); Bayer (Industry); Nuvation Bio Inc. (Industry); IQVIA Solutions Canada Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: CARMA-BROS; 18-5902 (Other: CAPCR-University Health Network); 1632 (Other: Clinical Trials Ontario (CTO)-Ontario Cancer Research Ethics Board (OCREB))
Record Dates: First submitted 2019-10-29; First posted 2019-11-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Malignancies Multiple; Malignant Solid Tumor; Cancer, Therapy-Related; Molecular Sequence Variation; Genetic Alteration; Gene Fusion; Receptor Tyrosine Kinase Gene Mutation; RTK Family Gene Mutation; Ras (Kras or Nras) Gene Mutation
Keywords: observational study; cancer; cancer therapies; molecular alterations; real-world evidence; real-world data; tyrosine kinase inhibitors; ambispective; ras GTPase inhibitors
MeSH Terms: conditions — Neoplasms; Neoplasms, Second Primary; Congenital Abnormalities | interventions — Tyrosine Kinase Inhibitors; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prospective: Living cancer patients with histologically confirmed rare molecular alterations in their tumours, such as in ALK, EGFR, ROS1, BRAF, and KRAS G12C from participating sites/cancer centres across Canada.
  Interventions: Drug: Cancer treatment with tyrosine kinase inhibitors (TKIs) or other molecularly targeted therapeutic agents.; Other: Patient-reported outcomes (PROs)
- Retrospective: Deceased cancer patients who had histologically confirmed rare molecular alterations in their tumours, such as in ALK, EGFR, ROS1, BRAF, and KRAS G12C from participating sites/cancer centres across Canada.
  Interventions: Drug: Cancer treatment with tyrosine kinase inhibitors (TKIs) or other molecularly targeted therapeutic agents.
- Comparator group: All cancer patients without rare molecular alterations in their solid tumours. This group will be established in order to determine baseline characteristics and outcomes, including treatment outcomes, of more standard treatments such as systemic chemotherapy or immunotherapy.

INTERVENTIONS:
Drug: Cancer treatment with tyrosine kinase inhibitors (TKIs) or other molecularly targeted therapeutic agents. — Observing cancer patients who have received or are currently receiving tyrosine kinase inhibitors (TKIs) or other molecularly targeted therapies for their cancer treatment.
  Groups: Prospective; Retrospective
Other: Patient-reported outcomes (PROs) — Prospectively enrolled participants will be provided with survey packets comprised of different PRO instruments at the initial/baseline visit, at 3 month follow up intervals and at the time when treatment/therapy is changed.
  Groups: Prospective

SUMMARY:
This study will collect data on Canadian cancer patients that have uncommon/rare changes in their tumours, such as alterations/rearrangements in the genetic material inside cells - known as deoxyribonucleic acid, or DNA, which acts as a map and gives directions to the cells on how to make other substances the body needs - because some of these changes have been found to respond to different drugs that help to stop the cancer. These rare changes occur in genes such as but not limited to ALK, EGFR, ROS1, BRAF, and NTRK which have targeted drugs in a family known as tyrosine kinase inhibitors (TKIs), and KRAS G12C mutation, which now has a targeted inhibitor drug therapy for patients with non small cell lung cancer (NSCLC). The goals for the study are to compare the natural history of such cancers and the treatment outcomes, including toxicities and patient-reported outcomes, for the different therapies.

DETAILED DESCRIPTION:
Molecular heterogeneity in cancer tumours make it a complex disease to manage and treat. However, there have been significant advancements made in the detection of molecular alterations and we are able to now define distinct disease subtypes which permit targeted selection of therapies, thus optimizing treatment responses for patients and improving their survival.

With CARMA-BROS we will address the objectives that follow.

Primary Objectives:

1. To create a cohort of patients through which to better understand the natural history of disease in Canadian cancer patients with tumours that have been molecularly subtyped and identified to have rare molecular alterations.
2. To compare the natural history, stage distribution, treatment outcomes such as treatment effectiveness (composite of disease progression or death) and treatment toxicities across different patients with different molecular alterations, receiving different lines and types of therapy.

   Secondary Objectives:
3. To determine the incidence, time to development, prevalence, and outcomes of patients with specific patterns of spread, such as brain metastases compared to those without, by different therapies and by molecular alterations.
4. To better understand real-world treatment patterns of rare molecular alterations in the Canadian context, across geographic or other factors, and how treatment patterns evolve over time and as new therapies become available, how patients are investigated and how targeted and other biomarkers are used as part of clinical practice in these patients.
5. To assess quality of life in patients with rare molecular alterations across different stages, lines and types of therapy.
6. To perform exploratory health economic evaluations focused on the costs and benefits of managing patients with rare molecular alterations.
7. To perform biomarker analyses, where appropriate, to improve our understanding of these rare molecular alterations.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years at cancer diagnosis
* Diagnosed with malignant tumour(s) with molecular testing completed that identified rare molecular alterations
* Accessible/available molecular testing reports/documentation to confirm type(s) of molecular alteration(s) (resulting from the conduct of polymerase chain reaction [PCR] based next generation sequencing [NGS], immunohistochemistry [IHC], fluorescence in situ hybridization [FISH], liquid biopsy)
* Canadian resident received follow-up for cancer care in Canada or is currently receiving/planning follow-up for cancer care to occur in Canada at time of enrollment

Exclusion Criteria:

* Previous refusal of the deceased patient, when living, to enroll in this study or patient approached for this study is unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients living and deceased who have/had a histologically confirmed rare molecular alteration in their tumours, such as but not limited to ALK, EGFR, ROS1, BRAF, and KRAS G12C from participating sites/cancer centres across Canada.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Composite of Progression Free Survival [PFS] or Overall Survival [OS] | From the start date of cancer therapy until the date of first documented progression or date of death (any cause), assessed up to 120 months
  Composite of disease progression or death

SECONDARY OUTCOMES:
Brain metastasis/other metastatic tumours | From the start date of cancer therapy until the date of first documented brain/other metastasis, assessed up to 120 months
  Confirmed through imaging (MRI, CT) or determined through treatment indication(s), for example, brain radiation therapy (surrogate for presence of brain metastasis)
EORTC quality of life questionnaires (QLQ) - cancer patient-reported health related quality of life | Baseline and serial changes every 3 months, including whenever there is a change in treatment, up to 120 months (the duration of this study)
  Prospectively enrolled participants will complete the following health related quality of life surveys: EORTC QLQ-C30 (core) and EORTC QLQ-LC13 (disease specific module)
EQ-5D-5L - patient-reported health related quality of life measure | Baseline and serial changes every 3 months, including whenever there is a change in treatment, up to 120 months (the duration of this study)
  Prospectively enrolled participants will complete the health related quality of life survey: EQ-5D-5L.
Patient-reported economic impact | Baseline and serial changes every 3 months, including whenever there is a change in treatment, up to 120 months (the duration of this study)
  Prospectively enrolled participants will complete the "Work Productivity and Activity Impairment Questionnaire: General Health" (WPAI:GH) and other economic impact questions that capture indirect costs incurred as a result of their disease.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Liu, MD, MSc, Principal Investigator — Princess Margaret Cancer Centre
Locations (27):
- Canada (27):
  - Tom Baker Cancer Centre - University of Calgary - Alberta Health Services, Calgary, Alberta
  - Cross Cancer Institute, University of Alberta - Alberta Health Services, Edmonton, Alberta
  - BC Cancer, Vancouver, British Columbia
  - CancerCare Manitoba/University of Manitoba, Winnipeg, Manitoba
  - Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II (QEII) Health Sciences Centre, Halifax, Nova Scotia
  - William Osler Health System - Brampton Civic Hospital, Brampton, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre (KHSC), Kingston, Ontario
  - Lawson Health Research Institute - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Princess Margaret Cancer Centre (PMCC) - University Health Network (UHN), Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Research Institute - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hôpital du Sacré-Coeur-de-Montréal (HSCM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Centre hospitalier de l'université de Québec - Université Laval, Québec, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided